CLINICAL TRIAL: NCT02129036
Title: Retrospective Multi-institutional Survey of Clinical Characteristics in Ovarian Clear Cell Adenocarcinoma Cancer Patients
Brief Title: Ovarian Clear Cell Adenocarcinoma Review
Acronym: OCCA
Status: Completed | Type: Observational
Sponsor: Cathay General Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ming Ho, Dr, Cathay General Hospital
Other Study IDs: TGOG-127
Record Dates: First submitted 2009-01-04; First posted 2014-05-02 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2014-04

CONDITIONS: Ovarian Cysts
Keywords: Ovarian cancer; Clear cell carcinoma; Paclitaxel-platinum; Chemotherapy; response to chemotherapy; survival of clear cell ovarian carcinoma; Prognostic factors
MeSH Terms: conditions — Ovarian Cysts; Ovarian Neoplasms; Adenocarcinoma, Clear Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clear cell carcinoma comprises 5-10% of surface epithelial ovarian cancers, and about 30-40% of the patients with clear cell carcinoma are diagnosed in the advanced stage. The investigators studied the response to chemotherapy and survival for either paclitaxel-platinum based chemotherapy or conventional platinum-based chemotherapy among all stages clear cell ovarian carcinoma. Prognostic factors for survival among the patients with pure, advanced, clear cell ovarian carcinoma were also evaluated.

DETAILED DESCRIPTION:
1. Several authors have reported frequent admixtures of clear cell ovarian carcinoma with serous, mucinous, and endometrioid tumors. However, few papers addressed the difference in response to chemotherapy and survival between patients with pure and mixed-type advanced clear cell carcinoma.
2. Recent trends in the clinical management of advanced ovarian cancer include increased attention to maximal cytoreduction and general acceptance of paclitaxel-platinum-based adjuvant chemotherapy.
3. The introduction of paclitaxel markedly changed the postoperative management of ovarian cancer patients, but the results and value of these newer efforts and therapies applied to clear cell carcinoma are as yet undetermined.
4. Today, paclitaxel-platinum-based chemotherapy is becoming the standard regimen for ovarian cancer worldwide. Previous research suggests a potential benefit of paclitaxel plus carboplatin regimens for stage I clear cell carcinoma. However, few papers specifically addressed the efficacy of paclitaxel-platinum-based chemotherapy for advanced clear cell carcinoma because clear cell carcinoma occurs only rarely in Western countries.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Ovarian clear cell carcinoma

Exclusion Criteria:

* not undergo operation

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: total 300 patients of ovarian clear cell carcinoma post operation from 8 institution.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Overall survival (up to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ming Ho, Study Director — Gynecologic Cancer Center, Cathay general Hospital